CLINICAL TRIAL: NCT01285674
Title: INTRATYMPANIC STEROID TREATMENT FOR THE PREVENTION OF INNER EAR TOXICITY ASSOCIATED WITH SYSTEMIC TREATMENT WITH CISPLATIN.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Dr Peter Gilbey, Ziv Medical Center, Safed, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0035-10-ZIV
Record Dates: First submitted 2011-01-23; First posted 2011-01-28 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Cisplatin; Ototoxicity; Intratympanic Steroids
Keywords: cisplatin; ototoxicity; intratympanic steroids
MeSH Terms: conditions — Ototoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra-tympanic steroid injection (Experimental)
  Interventions: Drug: Intra-tympanic Cisplatinum

INTERVENTIONS:
Drug: Intra-tympanic Cisplatinum — Intra-tympanic injection (under local anesthesia) of 0.5cc Methylprednisolone 62.5mg/cc. One injection per ear before each of the 3 cisplatin treatments. After injection the patient will remain with the treated ear upwards for 20 minutes and will try to avoid swallowing as much as possible.

SUMMARY:
In this study we will aim to determine if cisplatin ototoxicity can be prevented by intratympanic administration of corticosteroids.

DETAILED DESCRIPTION:
Cisplatin is a potent and widely used antineoplastic drug. Ototoxicity is a serious and dose-limiting side effect. The ototoxic effect of cisplatin is characterized by irreversible, progressive, bilateral, high-frequency, sensorineural hearing loss with tinnitus. 60-80% of patients treated show elevations of hearing thresholds and nearly 15% sustain significant hearing handicap. There are currently no clinical interventions that have been shown to prevent cisplatin ototoxicity in humans. Glucocorticoids have significant potential for otoprotection. Glucocorticoids are in use for treatment of a variety of cochlear disorders such as autoimmune inner ear disease, Meniere's disease and sudden sensorineural hearing loss. Intratympanic administration of drugs is a contemporary, safe method of locally treating inner ear disorders, allowing diffusion across the round window into the inner ear. This method achieves much higher steroid levels within the inner ear compared to oral or parenteral routes. Local administration prevents the common systemic side effects of steroids. Previous animal studies have shown protection against cisplatin-induced ototoxicity after intratympanic steroid injection. Asa far as we know, there are yet no studies in humans examining the otoprotective effect of intratympanic steroids in patients treated with cisplatin. In this study we will aim to determine if cisplatin ototoxicity can be prevented by intratympanic administration of corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years old at least who are candidates for Cisplatin treatment
* agreement to participate in the study
* have signed an informed consent.

Exclusion Criteria:

* refusal to participate
* steroid treatment during the past month
* external or middle ear disease not enabling intratympanic treatment
* inner ear disease causing hearing loss
* severe hearing loss for any reason
* conductive hearing loss

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Post-Treatment change in hearing | approximately 1 month from 1st treatment
  change in hearing as a result of cisplatin treatment as assessed by behavioural hearing test and otoacoustic emissions

SECONDARY OUTCOMES:
Tinnitus | 1 month post-treatment
  appearence or worsening of tinnitus as a result of cisplatin treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel